CLINICAL TRIAL: NCT04221789
Title: TB Treatment Support Tools: Refinement and Evaluation of an Interactive Mobile App and Direct Adherence Monitoring on TB Treatment Outcomes
Brief Title: TB Treatment Support Tool Interactive Mobile App and Direct Adherence Monitoring on TB Treatment Outcomes
Acronym: TB-TST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Effectiveness and Health Policy (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12112019
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis; Treatment Adherence
Keywords: treatment supervision, success default
MeSH Terms: conditions — Tuberculosis; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts will not be aware of group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention: TB treatment assistant (Experimental): Patients receiving instructions to use phone application
  Interventions: Other: TB treatment assistant
- Control (No Intervention): Patients receiving instructions for usual care self administered treatment

INTERVENTIONS:
Other: TB treatment assistant — Cell phone app to support self administered treatment and monitor adherence
  Other Names: TB-TST (Treatment Support Tools)
  Arms: intervention: TB treatment assistant

SUMMARY:
The overall goal of this study is to conduct a Randomized Clinical Trial (RCT) to evaluate a tuberculosis treatment support tool (TB-TST), a cellular phone app developed using user-centered design principles and a paper-based drug metabolite urine test strip modified for home use for testing the presence of isoniazid drug metabolites in urine to directly monitor adherence to treatment, to improve treatment outcomes for patients with TB receiving self-administered treatment (SAT).

Poor medication adherence to TB regimens, along with challenges in monitoring patients and returning them to treatment, are important contributing factors to poor outcomes and the development of drug resistance. With advances and proliferation of mobile technology platforms, there is substantial interest in the possible use of mobile health (mHealth) interventions to address these challenges. Of the mHealth approaches under investigation for TB adherence monitoring, drug metabolite testing has been identified as the most promising, ethical, and accurate, and the least intrusive and stigmatizing strategy compared to other mobile solutions, yet its potential remains largely unexplored. Additionally, mobile applications (apps) may provide personalized treatment supervision, increase patients' self-management and improve patient-provider communication by offering more advanced functionalities for patient support and monitoring.

The existing version of the TB-TST app offers education on TB and its treatment, communication with a care-coordinator, tracks treatment adherence (both by self-reporting and direct metabolite test strip images), self-reports treatment side-effects, and retains patient's "diary" notes. This proposal builds on preliminary work to: 1) Refine the TB-TST intervention based on pilot study findings and apply principles of user-centered design; 2) Evaluate the impact of the TB-TST on treatment outcomes compared to usual care; 3) Assess patient and provider perceptions of the facilitators and barriers to implementation of the TB-TST and synthesize lessons learned with stakeholders and policy makers. Primary outcome will be treatment success. Secondary outcomes will include: treatment default rates, self-reported adherence, technology use and usability. Findings have broader implications not only for TB adherence but disease management more generally and will improve our understanding of how to support patients facing challenging treatment regimens

DETAILED DESCRIPTION:
Tuberculosis remains one of the top ten causes of death globally despite it being largely curable. Patients face many challenges to adhere to treatment and mobile health (mHealth) interventions may address these challenges and support patients to complete their treatment. We will improve an interactive intervention based on the combined input from patients and TB experts and evaluate the intervention's impact on treatment outcomes in a randomized clinical trial. Findings have broader implications not only for TB adherence but disease management more generally and will improve our understanding of how to support patients in challenging treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 16 years old,
* have a new diagnosis of drug-susceptible TB,
* First treatment
* have regular access to a smartphone, and
* be able to operate the phone or have someone able to assist.

Exclusion Criteria:

* Children up to 15 years old
* Retreatment (default or previous treatment failure)
* Patients who are severely ill (i.e., requiring hospitalization)
* Patients who reside in the same household with another study participant
* Inability to operate a smartphone
* Illiteracy (inability to read and write)
* Patients with known drug resistance
* Patients with known HIV co-infection will be excluded because their care is managed separately.
* Screened patients who do not meet study eligibility will have specific screening data (including gender, age and reason for exclusion) entered into the study database to examine reasons for exclusion and feasibility of enrollment criteria.

Case definition: Patients at least 16 year old with TB confirmed by smear-positive sputum or diagnosis of pulmonary TB based on radiological findings and clinical signs and symptoms but with negative sputum smear. The diagnosis may be confirmed by other methods, such as, MGIT960, BACTEC 9000 or MB Bact, nucleic acid amplification (PCR) or ELISA.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando A Rubinstein, MD MPH, Principal Investigator — Institute for Clinical Effectiveness and Health Policy; Sarah Iribarren, RN PhD, Principal Investigator — University of Washington
Locations (1):
- IECS, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. The top 10 causes of death worldwide. Geneva, 2017.
- [Background] World Health Organization. Global Tuberculosis Report, 2018.
- [Background] World Health Organization. Tuberculosis: fact sheet no. 104, Reviewed March 2016, 2016.
- [Background] All Party Parliamentary Group on Global TB. The price of a pandemic:counting the cost of MDR-TB, 2015.
- [Background] World Health Organization. End TB Strategy. 2015.
- [Background] World Health Organization. Digital Health for the End TB Strategy: An Agenda for Action Geneva, Switzerland, 2015.
- [Background] World Health Organization. Digital health for the End TB strategy: progress since 2015 and future perspectives. Geneva: World Health Organization, 2017.
- [Background] DiStefano MJ, Schmidt H. mHealth for Tuberculosis Treatment Adherence: A Framework to Guide Ethical Planning, Implementation, and Evaluation. Glob Health Sci Pract. 2016 Jun 27;4(2):211-21. doi: 10.9745/GHSP-D-16-00018. Print 2016 Jun 20. PMID 27353615
- [Background] Schnall R, Bakken S, Brown Iii W, Carballo-Dieguez A, Iribarren S. Usabilty Evaluation of a Prototype Mobile App for Health Management for Persons Living with HIV. Stud Health Technol Inform. 2016;225:481-5. PMID 27332247
- [Background] Guerra RL, Conde MB, Efron A, Loredo C, Bastos G, Chaisson RE, Golub JE. Point-of-care Arkansas method for measuring adherence to treatment with isoniazid. Respir Med. 2010 May;104(5):754-7. doi: 10.1016/j.rmed.2010.02.001. Epub 2010 Mar 3. PMID 20202806
- [Background] Schraufnagel DE, Stoner R, Whiting E, Snukst-Torbeck G, Werhane MJ. Testing for isoniazid. An evaluation of the Arkansas method. Chest. 1990 Aug;98(2):314-6. doi: 10.1378/chest.98.2.314. PMID 2376164
- [Background] Kilburn JO, Beam RE, David HL, Sanchez E, Corpe RF, Dunn W. Reagent-impregnated paper strip for detection of metabolic products of isoniazid in urine. Am Rev Respir Dis. 1972 Dec;106(6):923-4. doi: 10.1164/arrd.1972.106.6.923. No abstract available. PMID 4641228
- [Background] World Health Organization. Global Tuberculosis Report, 2016. Geneva: World Health Organization, 2016.
- [Background] Fisher JD, Amico KR, Fisher WA, Harman JJ. The information-motivation-behavioral skills model of antiretroviral adherence and its applications. Curr HIV/AIDS Rep. 2008 Nov;5(4):193-203. doi: 10.1007/s11904-008-0028-y. PMID 18838059
- [Background] Schnall R, Rojas M, Bakken S, Brown W, Carballo-Dieguez A, Carry M, Gelaude D, Mosley JP, Travers J. A user-centered model for designing consumer mobile health (mHealth) applications (apps). J Biomed Inform. 2016 Apr;60:243-51. doi: 10.1016/j.jbi.2016.02.002. Epub 2016 Feb 20. PMID 26903153
- [Background] Center for Desease Control and Prevention. Tuberculosis Data and Statistics, 2018.
- [Background] Maartens G, Wilkinson RJ. Tuberculosis. Lancet. 2007 Dec 15;370(9604):2030-43. doi: 10.1016/S0140-6736(07)61262-8. PMID 17719083
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Ray TK, Sharma N, Singh MM, Ingle GK. Economic burden of tuberculosis in patients attending DOT centres in Delhi. J Commun Dis. 2005 Jun;37(2):93-8. PMID 16749271
- [Background] Corbett EL, Watt CJ, Walker N, Maher D, Williams BG, Raviglione MC, Dye C. The growing burden of tuberculosis: global trends and interactions with the HIV epidemic. Arch Intern Med. 2003 May 12;163(9):1009-21. doi: 10.1001/archinte.163.9.1009. PMID 12742798
- [Background] Iribarren SJ, Rubinstein F, Discacciati V, Pearce PF. Listening to Those at the Frontline: Patient and Healthcare Personnel Perspectives on Tuberculosis Treatment Barriers and Facilitators in High TB Burden Regions of Argentina. Tuberc Res Treat. 2014;2014:135823. doi: 10.1155/2014/135823. Epub 2014 Sep 28. PMID 25328701
- [Background] Hirpa S, Medhin G, Girma B, Melese M, Mekonen A, Suarez P, Ameni G. Determinants of multidrug-resistant tuberculosis in patients who underwent first-line treatment in Addis Ababa: a case control study. BMC Public Health. 2013 Aug 28;13:782. doi: 10.1186/1471-2458-13-782. PMID 23981845
- [Background] Mitchison DA. How drug resistance emerges as a result of poor compliance during short course chemotherapy for tuberculosis. Int J Tuberc Lung Dis. 1998 Jan;2(1):10-5. PMID 9562106
- [Background] Center for Desease Control and Prevention. The costly burden of drug-resistant TB in the U.S., 2017.
- [Background] World Health Organization. Global Plan to End TB: The Paradigm Shift 2016-2020. Geneva, Switzerland, 2015.
- [Background] World Health Organization. What is DOTS? A guide to understanding the WHO-recommended TB control strategy known as DOTS, 1999.
- [Background] Karumbi J, Garner P. Directly observed therapy for treating tuberculosis. Cochrane Database Syst Rev. 2015 May 29;2015(5):CD003343. doi: 10.1002/14651858.CD003343.pub4. PMID 26022367
- [Background] Pope DS, Chaisson RE. TB treatment: as simple as DOT? Int J Tuberc Lung Dis. 2003 Jul;7(7):611-5. PMID 12870680
- [Background] Volmink J, Garner P. Directly observed therapy for treating tuberculosis. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD003343. doi: 10.1002/14651858.CD003343.pub2. PMID 16625579
- [Background] Tuberculosis Coalition for Technical Assistance. International Standards for Tuberculosis Care (ISTC). Diagnosis, Treatment, Public Health. 2nd ed. The Hague, 2009.
- [Background] World Health Organization. Global Tuberculosis Report 2015. Geneva, Switzerland: WHO, 2015.
- [Background] Instituto Nacional de Enfermedades Respiratorias
- [Background] World Health Organization. TB country profile Argentina, 2017. 2018. http://www.who.int/tb/country/data/profiles/en/
- [Background] United Nations. Sustainable Development Goals. 2015. http://www.un.org/sustainabledevelopment/sustainable-development-goals/
- [Background] International telecommunication Union. The World in 2016: ICT Facts & Figures. 2016. http://www.itu.int/en/ITU-D/Statistics/Documents/facts/ICTFactsFigures2016.pdf
- [Background] Hoffman JA, Cunningham JR, Suleh AJ, Sundsmo A, Dekker D, Vago F, Munly K, Igonya EK, Hunt-Glassman J. Mobile direct observation treatment for tuberculosis patients: a technical feasibility pilot using mobile phones in Nairobi, Kenya. Am J Prev Med. 2010 Jul;39(1):78-80. doi: 10.1016/j.amepre.2010.02.018. Epub 2010 May 26. PMID 20537846
- [Background] Wade VA, Karnon J, Eliott JA, Hiller JE. Home videophones improve direct observation in tuberculosis treatment: a mixed methods evaluation. PLoS One. 2012;7(11):e50155. doi: 10.1371/journal.pone.0050155. Epub 2012 Nov 30. PMID 23226243
- [Background] Belknap R, Weis S, Brookens A, Au-Yeung KY, Moon G, DiCarlo L, Reves R. Feasibility of an ingestible sensor-based system for monitoring adherence to tuberculosis therapy. PLoS One. 2013;8(1):e53373. doi: 10.1371/journal.pone.0053373. Epub 2013 Jan 7. PMID 23308203
- [Background] Soobratty MR, Whitfield R, Subramaniam K, Grove G, Carver A, O'Donovan GV, Wu HH, Lee OY, Swaminathan R, Cope GF, Milburn HJ. Point-of-care urine test for assessing adherence to isoniazid treatment for tuberculosis. Eur Respir J. 2014 May;43(5):1519-22. doi: 10.1183/09031936.00132613. Epub 2014 Jan 16. No abstract available. PMID 24435008
- [Background] Singer E. TB Drug Compliance. Paper drug test and text messaging could help thwart the most deadly strains of tuberculosis. 2009. https://www.technologyreview.com/s/412203/tb-drug-compliance/
- [Background] Meissner PE, Musoke P, Okwera A, Bunn JE, Coulter JB. The value of urine testing for verifying adherence to anti-tuberculosis chemotherapy in children and adults in Uganda. Int J Tuberc Lung Dis. 2002 Oct;6(10):903-8. PMID 12365577
- [Background] Iribarren SJ, Sward KA, Beck SL, Pearce PF, Thurston D, Chirico C. Qualitative evaluation of a text messaging intervention to support patients with active tuberculosis: implementation considerations. JMIR Mhealth Uhealth. 2015 Feb 27;3(1):e21. doi: 10.2196/mhealth.3971. PMID 25802968
- [Background] Iribarren S, Beck S, Pearce PF, Chirico C, Etchevarria M, Cardinale D, Rubinstein F. TextTB: A Mixed Method Pilot Study Evaluating Acceptance, Feasibility, and Exploring Initial Efficacy of a Text Messaging Intervention to Support TB Treatment Adherence. Tuberc Res Treat. 2013;2013:349394. doi: 10.1155/2013/349394. Epub 2013 Dec 12. PMID 24455238
- [Background] Iribarren SJ, Beck SL, Pearce PF, Chirico C, Etchevarria M, Rubinstein F. MHEALTH INTERVENTION DEVELOPMENT TO SUPPORT PATIENTS WITH ACTIVE TUBERCULOSIS. J Mob Technol Med. 2014;3(2):16-27. doi: 10.7309/jmtm.3.2.4. PMID 26246859
- [Background] Rubinstein F, Iribarren, SJ. Effectiveness of different usual regimens treatment delivery strategies on Tuberculosis treatment success and default rates in Argentina: A Prospective Cohort Study (under review). 2017.
- [Background] Rubinstein F, Bernachea, M.P., Klein, K, Zurbrigk, F, Iribarren, S, Chirico, C, Gibbons, L,. TB treatment strategies and risk of default: a quasi-experimental study The International Journal of Tuberculosis and Lung Disease; 2016; Liverpool, UK; 2016.
- [Background] Fisher JD, Fisher WA, Amico KR, Harman JJ. An information-motivation-behavioral skills model of adherence to antiretroviral therapy. Health Psychol. 2006 Jul;25(4):462-73. doi: 10.1037/0278-6133.25.4.462. PMID 16846321
- [Background] Munro S, Lewin S, Swart T, Volmink J. A review of health behaviour theories: how useful are these for developing interventions to promote long-term medication adherence for TB and HIV/AIDS? BMC Public Health. 2007 Jun 11;7:104. doi: 10.1186/1471-2458-7-104. PMID 17561997
- [Background] McReynolds J, Crane, H, Berry, D, Lober, WB. Open Source Computerized Patient Reported Outcomes: Research and Practice across Three Domains. AMIA; 2013; Washington DC; 2013.
- [Background] Mandel JC, Kreda DA, Mandl KD, Kohane IS, Ramoni RB. SMART on FHIR: a standards-based, interoperable apps platform for electronic health records. J Am Med Inform Assoc. 2016 Sep;23(5):899-908. doi: 10.1093/jamia/ocv189. Epub 2016 Feb 17. PMID 26911829
- [Background] Banos O, Villalonga C, Garcia R, Saez A, Damas M, Holgado-Terriza JA, Lee S, Pomares H, Rojas I. Design, implementation and validation of a novel open framework for agile development of mobile health applications. Biomed Eng Online. 2015;14 Suppl 2(Suppl 2):S6. doi: 10.1186/1475-925X-14-S2-S6. Epub 2015 Aug 13. PMID 26329639
- [Background] Flood D, Chary A, Austad K, Diaz AK, Garcia P, Martinez B, Canu WL, Rohloff P. Insights into Global Health Practice from the Agile Software Development Movement. Glob Health Action. 2016 Apr 29;9:29836. doi: 10.3402/gha.v9.29836. eCollection 2016. PMID 27134081
- [Background] Ngwatu BK, Nsengiyumva NP, Oxlade O, Mappin-Kasirer B, Nguyen NL, Jaramillo E, Falzon D, Schwartzman K; Collaborative group on the impact of digital technologies on TB. The impact of digital health technologies on tuberculosis treatment: a systematic review. Eur Respir J. 2018 Jan 11;51(1):1701596. doi: 10.1183/13993003.01596-2017. Print 2018 Jan. PMID 29326332
- [Background] Alipanah N, Jarlsberg L, Miller C, Linh NN, Falzon D, Jaramillo E, Nahid P. Adherence interventions and outcomes of tuberculosis treatment: A systematic review and meta-analysis of trials and observational studies. PLoS Med. 2018 Jul 3;15(7):e1002595. doi: 10.1371/journal.pmed.1002595. eCollection 2018 Jul. PMID 29969463
- [Background] Iribarren S, Schnall R. Call for Increased Patient Support Focus: Review and Evaluation of Mobile Apps for Tuberculosis Prevention and Treatment. Stud Health Technol Inform. 2016;225:936-7. PMID 27332418
- [Background] eMarketer. Smartphone uptake is on the rise in Argentina. 4G is becoming more common. Aug 4, 2016 2016. https://www.emarketer.com/Article/Smartphone-Uptake-on-Rise-Argentina/1014300 (accessed Aug 17 2018).
- [Background] Atun R, Weil DE, Eang MT, Mwakyusa D. Health-system strengthening and tuberculosis control. Lancet. 2010 Jun 19;375(9732):2169-78. doi: 10.1016/S0140-6736(10)60493-X. Epub 2010 May 18. PMID 20488514
- [Background] Lonnroth K, Jaramillo E, Williams BG, Dye C, Raviglione M. Drivers of tuberculosis epidemics: the role of risk factors and social determinants. Soc Sci Med. 2009 Jun;68(12):2240-6. doi: 10.1016/j.socscimed.2009.03.041. Epub 2009 Apr 23. PMID 19394122
- [Background] Volpp K. A healthcare revolution: Behavioral economics for behavior change and preventive medicine. NIH Office of Behavioral and Social Sciences Research; 2015.
- [Background] Masterson Creber RM, Maurer MS, Reading M, Hiraldo G, Hickey KT, Iribarren S. Review and Analysis of Existing Mobile Phone Apps to Support Heart Failure Symptom Monitoring and Self-Care Management Using the Mobile Application Rating Scale (MARS). JMIR Mhealth Uhealth. 2016 Jun 14;4(2):e74. doi: 10.2196/mhealth.5882. PMID 27302310
- [Background] Berry DL, Hong F, Halpenny B, Partridge A, Fox E, Fann JR, Wolpin S, Lober WB, Bush N, Parvathaneni U, Amtmann D, Ford R. The electronic self report assessment and intervention for cancer: promoting patient verbal reporting of symptom and quality of life issues in a randomized controlled trial. BMC Cancer. 2014 Jul 12;14:513. doi: 10.1186/1471-2407-14-513. PMID 25014995
- [Background] Evans HL, Lober WB. A Pilot Use of Patient-Generated Wound Data to Improve Postdischarge Surgical Site Infection Monitoring. JAMA Surg. 2017 Jun 1;152(6):595-596. doi: 10.1001/jamasurg.2017.0568. No abstract available. PMID 28423162
- [Background] Fredericksen RJ, Tufano J, Ralston J, McReynolds J, Stewart M, Lober WB, Mayer KH, Mathews WC, Mugavero MJ, Crane PK, Crane HM. Provider perceptions of the value of same-day, electronic patient-reported measures for use in clinical HIV care. AIDS Care. 2016 Nov;28(11):1428-33. doi: 10.1080/09540121.2016.1189501. Epub 2016 May 29. PMID 27237187
- [Background] Chirico C, Kuriger A, Etchevarria M, Casamajor L, Morcillo N. Is the DOTS strategy a useful tool to fight against Tuberculosis in a median incidence area of Buenos Aires Province? Int J Tuberc Lung Dis 2005.
- [Background] Chirico C, Kuriger A, Fernandez H, Morcillo N. [Tuberculosis in the V Sanitary Zone of Buenos Aires Province. Analysis of its trends between 1984 and 1996]. Medicina (B Aires). 1999;59(4):332-8. Spanish. PMID 10752196
- [Background] Chirico C, Sanjurjo M, Iribarren S, Appendino A, Zerbini E, Etchevarria M. [Trends of tuberculosis in the Fifth Health Region, Buenos Aires Province, years 2000-2011]. Medicina (B Aires). 2015;75(3):147-54. Spanish. PMID 26117604
- [Background] mPOWEr - University of Washington. mPOWEr. 2016. http://mpowercare.org/ (accessed Sept 4 2016).
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Zelenko O, Tjondronegoro D, Mani M. Mobile app rating scale: a new tool for assessing the quality of health mobile apps. JMIR Mhealth Uhealth. 2015 Mar 11;3(1):e27. doi: 10.2196/mhealth.3422. PMID 25760773
- [Background] Akraa S, Tran Tama, A, Shena, H, Tang, Y, Tang, B.Z, Li, J, Walker, S. A smartphone-based point-of-care quantitative urinalysis device for chronic kidney disease patients. Journal of Network and Computer Applications 2018; 115(2018): 59-69.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Statista. Smartphone users as share of the population in Argentina from 2015 to 2022. 2018. https://www.statista.com/statistics/621034/smartphone-user-penetration-in-argentina/
- [Background] Instituto Nacional de Enfermedades Respiratorias. Programa Nacional de Control de la tuberculosis. Normas tecnicas (National Tuberculosis Program. Technical standards), 2002.
- [Background] Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, Kindelan JM, Carmona A, Juega J, Ocampo A; GEEMA Study Group. Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. AIDS. 2002 Mar 8;16(4):605-13. doi: 10.1097/00002030-200203080-00012. PMID 11873004
- [Background] Treatment of Tuberculosis: Guidelines. 4th edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138748/ PMID 23741786
- [Background] Guest G, Namey, E, Taylor, J, Eley, N & McKenna, K. Comparing focus groups and individual interviews: findings from a randomized study. International Journal of Social Research Methodology 2017; 20(6): 693-708.
- [Background] Mani M, Kavanagh DJ, Hides L, Stoyanov SR. Review and Evaluation of Mindfulness-Based iPhone Apps. JMIR Mhealth Uhealth. 2015 Aug 19;3(3):e82. doi: 10.2196/mhealth.4328. PMID 26290327
- [Background] Lincoln Y, Guba E. Naturalistic Inquiry. Newbury Park, CA: Sage Publications; 1985.
- [Background] Creswell JW, Klassen, A. C., Plano-Clark, V. L., Smith, K. C., for Office of Behavioral and Social Sciences Research. Best practices for mixed method research in the health sciences. Washington, DC: NIH National Institutes of Health, 2011.
- [Background] Johnson RB, Onwuegbuzie AJ. Mixed methods research: A research paradigm whose time has come Educational Researcher 2004; 33(7): 14-26.
- [Background] Thomas DR. A General Inductive Approach for Analyzing Qualitative Evaluation Data. American Journal of Evaluation 2006; 27(2): 237-46.
- [Derived] Roberti J, Morelli DM, Aguilar-Vidrio OA, Suyanto A, Carmiol-Rodriguez P, Tolentino A, Chen-Liang E, Sprecher J, Rubinstein F, Iribarren S. Improving tuberculosis treatment adherence: a qualitative study of patients' perspectives from a pragmatic trial of the tuberculosis treatment support tools intervention. BMJ Open. 2025 Sep 2;15(9):e095878. doi: 10.1136/bmjopen-2024-095878. PMID 40897502
- [Derived] Iribarren S, Milligan H, Goodwin K, Aguilar Vidrio OA, Chirico C, Telles H, Morelli D, Lutz B, Sprecher J, Rubinstein F. Mobile Tuberculosis Treatment Support Tools to Increase Treatment Success in Patients with Tuberculosis in Argentina: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jun 21;10(6):e28094. doi: 10.2196/28094. PMID 34152281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2020 and May 2023, a total of 555 individuals were enrolled across four public reference hospitals in Argentina. Of the 1017 individuals assessed for eligibility, 380 were excluded mostly due to retreatment
Period: Overall Study
Arm/Group | Intervention: TB Treatment Assistant | Control
Started | 277 | 278
Completed | 255 | 270
Not Completed | 22 | 8
Not completed — deviation from protoco | 22 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: TB Treatment Assistant | Control | Total
Number analyzed (Participants) | 277 | 278 | 555
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (12.97) | 33.7 (13.66) | 33.1 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 135 | 280
  Male | 132 | 143 | 275
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success
Description: Number of participants who completed 6 months of treatment and/ or demonstrated a bacteriological cure after 6 months
Time Frame: 6 months
Population: No differences
Measure: Number; unit: Participants
Arm/Group | Intervention: TB Treatment Assistant | Control
Number analyzed (Participants) | 255 | 270
Participants | 208 | 201
Statistical Analysis 1: Comparison: Intervention: TB Treatment Assistant vs Control; Ho no difference in treatment success between groups. The study was originally powered to detect a 15% difference between groups; Test type: Other — differences in proportions; p = 0.049, Chi-squared — Statistical significance threshold p <0.05; Risk Ratio (RR) = 1.12, 95% CI 2-sided [1.02 to 1.20]

2. Secondary Outcome: Treatment Default
Description: Abandonment of treatment for at least 2 months
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Intervention: TB Treatment Assistant | Control
Number analyzed (Participants) | 255 | 270
Participants | 44 | 66
Statistical Analysis 1: Comparison: Intervention: TB Treatment Assistant vs Control; Ho No difference between arms. 80% power to detect a 10% difference; Test type: Other — comparison of proportions and relative risk with 95% CI; p < 0.043, Chi-squared — statistical significance if p value <0.05; Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.50 to 0.97] — intervention / control

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention: TB Treatment Assistant | Control
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/278
Serious Adverse Events (participants affected / at risk) | 0/277 | 0/278
Other Adverse Events (participants affected / at risk) | 0/277 | 0/278

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04221789/Prot_SAP_000.pdf